CLINICAL TRIAL: NCT00762346
Title: Efficacy and Safety Study of ZOMETA® in Treatment of High-level NTX Non Small Cell Lung Cancer With Bone Metastasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446ECN06T
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2011-12

CONDITIONS: Non Small Cell Lung Cancer; Bone Metastases; High NTX Level
Keywords: non small cell lung cancer; NTX; zometa
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: zometa

INTERVENTIONS:
Drug: zometa — zometa 4mg i.v. every 4 weeks for up to 2 years

SUMMARY:
A multicenter prospective study to assess the efficacy and safety of ZOMETA® in treatment of high-level NTX non small cell lung cancer with bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically confirmed non-small cell cancer
* One bone metastasis at least confirmed by image(X ray, CT or others)
* NTX > 50nM BCE/mM creatinine
* Life expectancy > 6 M
* ECOG <= 2
* Signed ICF

Exclusion Criteria:

* Women who are pregnant or in lactation
* Patients with hyperostosis with brain metastasis(exception of those without symptom or with Metastasis Lesions under controlled
* Previous or current treatment with any other bisphosphonates, bone- protecting, cytotoxic or targeted therapy
* Severe co-morbidity of any type that may interfere with assessment of the patient for the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Skeleton-related event | 2 years

SECONDARY OUTCOMES:
OS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- cancer center, Sun Yat-sen University, Guangzhou, Guangdong, China